CLINICAL TRIAL: NCT07234786
Title: Prospective, Multicentric, Single Arm Clinical Investigation to Assess the Effectiveness and Safety of Multi-Gyn FemiTotal for Treatment and Prevention of Vulvovaginal Candidiasis Symptoms and Bacterial Vaginosis.
Brief Title: Clinical Study of a Vaginal Gel for the Treatment and Prevention of Vaginal Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-1774-U5 / 24INSE105
Record Dates: First submitted 2025-09-25; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Bacterial Vaginosis; Vaginal Candidiasis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal

STUDY DESIGN:
Intervention Model Description: Vaginal gel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study product (Experimental): Multi-Gyn Femitotal vaginal gel
  Interventions: Device: Multi-Gyn FemiTotal

INTERVENTIONS:
Device: Multi-Gyn FemiTotal — vaginal gel

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of Multi-Gyn Femitotal to treat and prevent women suffering from bacterial vaginosis and vulvo vaginal candidiasis. 40 subjects with itching symptoms of VVC and 49 subjects with BV as confirmed using Amsel criteria will be included and will use the device for 7 days (treatment phase). If the VVC symptoms and BV are considered as cured 21 days after the beginning of treatment, the subjects will be followed-up until Month 4 after treatment initiation to check the re-occurrence of VVC and BV (prevention phase).The primary objective is to evaluate the effectiveness of Multi-Gyn FemiTotal for the treatment of Bacterial Vaginosis (BV) and relief of VulvoVaginal Candidiasis (VVC) itching, 21 days after treatment initiation.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old.
2. Women suffering from VVC or BV at the time of inclusion:
3. For VVC: Subject with at least itching score > 2 and crumbly white discharge.
4. For BV: Subject with at least 3 out of 4 Amsel criteria positive, with at least presence of clue cells (>20%).

   Amsel criteria used for the study:
   * Thin, white, yellow, homogeneous discharge,
   * Clue cells on wet mount microscopy >20%,
   * a vaginal fluid pH ≥4.5 when placing the discharge on litmus paper,
   * Release fishy odor after adding 10% potassium hydroxide (KOH) solution to wet mount - also known as "whiff test".
5. Subject having given freely and expressly her informed consent.
6. Subject using a contraceptive regimen recognized as effective (pill, implant, Intra Uterine Device (IUD), condoms) since at least 12 weeks before inclusion visit and during the whole study.
7. Subject cooperative and aware of the device's modalities of use and the necessity and duration of the follow-up visits so that perfect adhesion to the protocol can be expected

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject suspected to be non-compliant according to the investigator's judgment.
3. Subject enrolled in another clinical trial during the study period on the vaginal area.
4. Subject having a known allergy or hypersensitivity to one of the components of the investigational device.
5. Subject suffering from a sexually transmitted gynaecological infection, genital tract infection or aerobic vaginitis (including clinical obvious gonorrhoea, chlamydia trachomatis or mycoplasma genitalium infection with cervicitis, urethritis, salpingitis).
6. Subject with current genital malignancies.
7. Subject who had a chemotherapy treatment in the 6 months before inclusion.
8. Subject who had a radiotherapy treatment in the genito-urinary area in the 12 months before inclusion.
9. Subject using treatment for vaginal conditions, vaginal infections, or other intravaginal treatment at the time of inclusion.
10. Subject using antibiotics for any reason in the 14 days before inclusion.
11. Subject using vaginal douches and who do not wish to refrain using them during the clinical investigation.
12. Subject with a pessary.
13. Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only
Enrollment: 80 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of Multi-Gyn FemiTotal for the treatment of Bacterial Vaginosis (BV) and relief of VulvoVaginal candidiasis symptoms will be evaluated by the investigator and questionnaires. | 21 days
  Cured rated of subjects with BV will be evaluated based on Amsel criteria. Subjects with VVC will be evaluated based on improvement of the itch.

SECONDARY OUTCOMES:
The prevention of BV and VVC re-occurrence will be evaluated by the doctor, 4 months after using the product. | 4 months
  Percentage of subjects without relapse of BV or VVC, 4 months after treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Farah Bolaky, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No